CLINICAL TRIAL: NCT01033201
Title: The Role Of Endoscopic Alveoscopy by Confocal Endomicroscopy in Diagnosing Acute and Chronic Rejection in Lung Transplant Recipients, Diagnosis of End Stage Lung Disease, and Other Pulmonary Pathologies in Vivo
Brief Title: Alveoscopy, Endoscopic Confocal Microscopy and Lung Rejection, Parenchymal Lung Diseases in Vivo
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Cesar A. Keller, M.D., Mayo Clinic Florida
Other Study IDs: 08-000800; ACA00001534
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Lung Transplant
Keywords: Lung rejection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung transplant: All lung transplant patients presenting for screening/surveillance and diagnostic bronchoscopies at Mayo Clinic Florida are eligible for participation.
  Interventions: Other: Confocal imaging

INTERVENTIONS:
Other: Confocal imaging — At the time of the standard of care bronchoscopy, confocal images will be obtained from each consented patient.
  Other Names: AlveoloFlex Confocal Miniprobes; Cellvizio-Lung system

SUMMARY:
Lung transplantation is indicated when end-stage lung diseases no longer respond to available standard therapy, making life expectancy short and associated with disability. Acute and chronic rejection are common complications following transplantation, indicating screening bronchoscopies and transbronchial biopsies at three month intervals the first two years, in addition to clinically indicated procedures when rejection or infection is suspected. Transbronchial biopsies carry associated risks (bleeding, pneumothorax). Chronic rejection is characterized by progressive obliteration of distal airways (Bronchiolitis Obliterans-BO-). BO requires open lung biopsy for diagnosis. Alternatively, a clinical surrogate (Bronchiolitis Obliterans Syndrome), characterized by decline in Forced Expired Volume in 1 second not explained by acute rejection or infection is used for diagnosis. The new technique of confocal endo-microscopy enables sub-surface visualization of tissue in vivo during bronchoscopic procedures using a probe-based confocal microscope, integrated to a standard endoscope. Bronchiolar and alveolar structures can be visualized at a cellular and nuclear level, and these images can be saved and reviewed. This new technology could potentially identify acute and chronic rejection, thus offering and alternative to transbronchial biopsies. We expect to describe a new alternative to diagnose acute and chronic rejection using confocal microscopy images obtained endoscopically, obviating complications of transbronchial biopsies.

Endoscopic confocal endomicroscopy can detect and classify common bronchiolar and alveolar pathological conditions in real time. Specifically, we hypothesize that confocal endomicroscopy images of bronchiolar and alveolar structures during standard bronchoscopy could help to recognize and classify the presence/absence of acute rejection and/or bronchiolitis obliterans syndrome in lung transplant recipients. This technology could also identify the histological characteristics lung diseases such as interstitial, obstructive or vascular end stage lung diseases, and thus lead to more efficient, safer and more accurate diagnosis of these lung conditions during routine bronchoscopies.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Any patient undergoing surveillance or clinically indicated bronchoscopies during or after lung transplantation
3. Any patient undergoing bronchoscopy prior lung transplant

Exclusion Criteria:

1. Unwilling to consent
2. Unable to safely tolerate a bronchoscopic procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo bronchoscopy either before or after lung transplantation.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2008-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine in an unblinded study, the key image features of acute lung rejection and chronic lung rejection (BOS), and estimate which morphologic features best distinguish these conditions. | One year

SECONDARY OUTCOMES:
To determine the initial sensitivity and specificity of confocal imaging for the classification of acute lung rejection among lung transplant recipients. | One year
To develop a library of confocal images with the most optimal confocal imaging characteristics of other lung pathologies requiring lung transplantation. | One year
To determine the inter-examiner differences and learning curve for accurate detection of acute rejection as well as the confocal images of other lung pathologies. | One year
To determine in a unblinded pilot study, the key image features of chronic lung rejection as defined by the Bronchiolitis Obliterans Syndrome (BOS), and estimate which morphologic features best distinguish this conditions. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- [Background] St Croix CM, Leelavanichkul K, Watkins SC. Intravital fluorescence microscopy in pulmonary research. Adv Drug Deliv Rev. 2006 Sep 15;58(7):834-40. doi: 10.1016/j.addr.2006.07.007. Epub 2006 Aug 11. PMID 16996641
- [Background] Herth FJ, Eberhardt R, Ernst A. The future of bronchoscopy in diagnosing, staging and treatment of lung cancer. Respiration. 2006;73(4):399-409. doi: 10.1159/000093369. PMID 16775411
- [Background] Trulock EP, Christie JD, Edwards LB, Boucek MM, Aurora P, Taylor DO, Dobbels F, Rahmel AO, Keck BM, Hertz MI. Registry of the International Society for Heart and Lung Transplantation: twenty-fourth official adult lung and heart-lung transplantation report-2007. J Heart Lung Transplant. 2007 Aug;26(8):782-95. doi: 10.1016/j.healun.2007.06.003. No abstract available. PMID 17692782
- [Background] Moffatt SD, Demers P, Robbins RC, Doyle R, Wienacker A, Henig N, Theodore J, Reitz BA, Whyte RI. Lung transplantation: a decade of experience. J Heart Lung Transplant. 2005 Feb;24(2):145-51. doi: 10.1016/j.healun.2003.10.020. PMID 15701428
- [Background] Sibley RK, Berry GJ, Tazelaar HD, Kraemer MR, Theodore J, Marshall SE, Billingham ME, Starnes VA. The role of transbronchial biopsies in the management of lung transplant recipients. J Heart Lung Transplant. 1993 Mar-Apr;12(2):308-24. PMID 8476904
- [Background] Bowdish ME, Arcasoy SM, Wilt JS, Conte JV, Davis RD, Garrity ER, Hertz ML, Orens JB, Rosengard BR, Barr ML. Surrogate markers and risk factors for chronic lung allograft dysfunction. Am J Transplant. 2004 Jul;4(7):1171-8. doi: 10.1111/j.1600-6143.2004.00483.x. PMID 15196078
- [Background] Colombat M, Groussard O, Lautrette A, Thabut G, Marrash-Chahla R, Brugiere O, Mal H, Leseche G, Fournier M, Degott C. Analysis of the different histologic lesions observed in transbronchial biopsy for the diagnosis of acute rejection. Clinicopathologic correlations during the first 6 months after lung transplantation. Hum Pathol. 2005 Apr;36(4):387-94. doi: 10.1016/j.humpath.2005.01.022. PMID 15892000
- [Background] Khalifah AP, Hachem RR, Chakinala MM, Yusen RD, Aloush A, Patterson GA, Mohanakumar T, Trulock EP, Walter MJ. Minimal acute rejection after lung transplantation: a risk for bronchiolitis obliterans syndrome. Am J Transplant. 2005 Aug;5(8):2022-30. doi: 10.1111/j.1600-6143.2005.00953.x. PMID 15996255
- [Background] Hachem RR, Yusen RD, Chakinala MM, Meyers BF, Lynch JP, Aloush AA, Patterson GA, Trulock EP. A randomized controlled trial of tacrolimus versus cyclosporine after lung transplantation. J Heart Lung Transplant. 2007 Oct;26(10):1012-8. doi: 10.1016/j.healun.2007.07.027. PMID 17919621
- [Background] Tazelaar HD, Nilsson FN, Rinaldi M, Murtaugh P, McDougall JC, McGregor CG. The sensitivity of transbronchial biopsy for the diagnosis of acute lung rejection. J Thorac Cardiovasc Surg. 1993 Apr;105(4):674-8. PMID 8469001
- [Background] Yousem SA, Berry GJ, Cagle PT, Chamberlain D, Husain AN, Hruban RH, Marchevsky A, Ohori NP, Ritter J, Stewart S, Tazelaar HD. Revision of the 1990 working formulation for the classification of pulmonary allograft rejection: Lung Rejection Study Group. J Heart Lung Transplant. 1996 Jan;15(1 Pt 1):1-15. PMID 8820078
- [Background] Estenne M, Maurer JR, Boehler A, Egan JJ, Frost A, Hertz M, Mallory GB, Snell GI, Yousem S. Bronchiolitis obliterans syndrome 2001: an update of the diagnostic criteria. J Heart Lung Transplant. 2002 Mar;21(3):297-310. doi: 10.1016/s1053-2498(02)00398-4. No abstract available. PMID 11897517
- [Background] Kiesslich R, Burg J, Vieth M, Gnaendiger J, Enders M, Delaney P, Polglase A, McLaren W, Janell D, Thomas S, Nafe B, Galle PR, Neurath MF. Confocal laser endoscopy for diagnosing intraepithelial neoplasias and colorectal cancer in vivo. Gastroenterology. 2004 Sep;127(3):706-13. doi: 10.1053/j.gastro.2004.06.050. PMID 15362025
- [Background] Thiberville L, Moreno-Swirc S, Vercauteren T, Peltier E, Cave C, Bourg Heckly G. In vivo imaging of the bronchial wall microstructure using fibered confocal fluorescence microscopy. Am J Respir Crit Care Med. 2007 Jan 1;175(1):22-31. doi: 10.1164/rccm.200605-684OC. Epub 2006 Oct 5. PMID 17023733
- [Background] Pacurariu RI. Low incidence of side effects following intravenous fluorescein angiography. Ann Ophthalmol. 1982 Jan;14(1):32-6. PMID 7125438